CLINICAL TRIAL: NCT07351396
Title: THE EFFECT OF VOLLEYBALL-SPECIFIC INJURY PREVENTION PROGRAM ON DYNAMIC BALANCE AND POSTURAL STABILITY IN YOUNG MALE VOLLEYBALL PLAYERS: A RANDOMIZED CONTROLLED TRIAL
Brief Title: The Effect of Volleyball-Specific Injury Prevention Program on Dynamic Balance and Postural Stability in Young Male Volleyball Players; Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Salih PINAR, Salih PINAR, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 57.2023FBU
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Healthy Adult Male; Volleyball Players; Injury Prevention in Sports; Neuromuscular Performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VOLLEY12+ Group (Experimental): Participants performed a progressive volleyball-specific neuromuscular warm-up program (VOLLEY 12+) before each training session for 12 weeks. The program lasted 16-20 minutes and included dynamic mobility, balance, landing mechanics, trunk and hip control, and shoulder activation exercises.
  Interventions: Other: VOLLEY12+ Volleyball-Specific Warm-Up Program
- Control Group (Active Comparator): Participants performed their usual coach-led warm-up routines before each training session for 12 weeks. The routine included low-intensity jogging, dynamic mobility and stretching exercises, and volleyball-specific ball-handling activities, without any structured neuromuscular or injury-prevention content.
  Interventions: Other: Regular Coach-Led Volleyball Warm-Up

INTERVENTIONS:
Other: Regular Coach-Led Volleyball Warm-Up — Participants performed their usual coach-led warm-up routine prior to volleyball training. This routine consisted of low-intensity jogging, dynamic mobility, and stretching exercises, followed by basic volleyball-specific ball-handling drills. No structured injury-prevention or neuromuscular training components were included, and the content was not modified by the research team.
  Arms: Control Group
Other: VOLLEY12+ Volleyball-Specific Warm-Up Program — A progressive volleyball-specific neuromuscular warm-up program (VOLLEY12+) performed before regular training sessions over a 12-week period. The program was designed to enhance dynamic balance, neuromuscular control, and landing mechanics by targeting the ankle, knee, hip, and shoulder regions. Exercises were progressively overloaded using changes in volume, distance, and external resistance, and the total duration of each session was approximately 16-20 minutes.
  Arms: VOLLEY12+ Group

SUMMARY:
The purpose of this study is to examine the effects of a 12-week volleyball-specific warm-up program (VOLLEY12+) on neuromuscular performance in young male volleyball players. Neuromuscular performance is an important factor related to injury risk and athletic performance in youth sports.

Twenty-four male volleyball players aged 15 to 17 years were allocated into an intervention group or a control group. The intervention group performed the VOLLEY12+ warm-up program before each training session for 12 weeks, while the control group continued their usual coach-led warm-up routines. Neuromuscular performance was assessed before and after the intervention using balance and movement control tests, including the Balance Error Scoring System (BESS), the Landing Error Scoring System (LESS), and the Y Balance Test.

The results of this study will help determine whether a structured, sport-specific warm-up program can improve neuromuscular performance in adolescent volleyball players and support the use of injury prevention strategies in youth volleyball training.

ELIGIBILITY:
Inclusion Criteria:

* Male volleyball players aged 15-17 years
* At least 3 years of volleyball training experience
* Regular volleyball training ≥3 days per week, ≥60 minutes per session
* No history of chronic or recurrent injury
* Voluntary participation with informed consent

Exclusion Criteria:

* Injury occurring during the study period
* Voluntary withdrawal from the study
* Inability to continue participation due to injury during the research process

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Static Balance Performance Assessed by the Balance Error Scoring System (BESS) | Baseline and after 12 weeks
  Static balance performance was assessed using the Balance Error Scoring System (BESS). Participants performed double-leg, single-leg, and tandem stances on firm and foam surfaces. Each stance was held for 20 seconds, and balance errors were recorded by a blinded assessor. Total error scores were calculated at baseline (pre-intervention) and after the 12-week intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahçe Sports Club - Dereağzı Facilities, Volleyball Hall, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bere T, Kruczynski J, Veintimilla N, Hamu Y, Bahr R. Injury risk is low among world-class volleyball players: 4-year data from the FIVB Injury Surveillance System. Br J Sports Med. 2015 Sep;49(17):1132-7. doi: 10.1136/bjsports-2015-094959. Epub 2015 Jul 20. PMID 26194501
- [Background] de Azevedo Sodre Silva A, Sassi LB, Martins TB, de Menezes FS, Migliorini F, Maffulli N, Okubo R. Epidemiology of injuries in young volleyball athletes: a systematic review. J Orthop Surg Res. 2023 Oct 4;18(1):748. doi: 10.1186/s13018-023-04224-3. PMID 37789463
- [Background] Zarei M, Eshghi S, Hosseinzadeh M. The effect of a shoulder injury prevention programme on proprioception and dynamic stability of young volleyball players; a randomized controlled trial. BMC Sports Sci Med Rehabil. 2021 Jun 30;13(1):71. doi: 10.1186/s13102-021-00300-5. PMID 34193267
- [Background] Verhagen E, Vriend I, Gouttebarge V, Kemler E, de Wit J, Zomerdijk D, Nauta J. Effectiveness of a warm-up programme to reduce injuries in youth volleyball players: a quasi-experiment. Br J Sports Med. 2023 Apr;57(8):464-470. doi: 10.1136/bjsports-2022-105425. Epub 2023 Feb 17. PMID 36801807